CLINICAL TRIAL: NCT01650493
Title: In-situ Evaluation of Anti-caries Technology
Status: Completed | Type: Observational
Sponsor: Solventum US LLC (Industry)
Collaborators: University of Iowa (Other); 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-11-012
Record Dates: First submitted 2012-06-14; First posted 2012-07-26 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Caries
Keywords: remineralization; demineralzation; in situ; dentrifice

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Clinpro 5000
  Interventions: Device: Clinpro 5000
- Group B: MI Paste Plus
  Interventions: Device: MI Paste Plus
- Group C: Toms of Maine
  Interventions: Device: Tom's of Maine

INTERVENTIONS:
Device: Clinpro 5000 — Dentrifice containing 950ppm fluoride
  Groups: Group A
Device: MI Paste Plus — Dentrifice containing 950ppm fluoride
  Groups: Group B
Device: Tom's of Maine — Dentrifice that is fluoride free
  Groups: Group C

SUMMARY:
Three toothpastes will be compared, two toothpastes in each subject, to establish whether changes in the depth or area of an artificially created area of tooth decay is the same for each toothpaste.

DETAILED DESCRIPTION:
Objective is to evaluate the demineralization and remineralization effects of two experimental fluoride containing dentrifices on enamel and root surface lesions compared with a control dentrifice.

Study is a partially randomized, 3-period cross over study involving 30 subjects who need a full-coverage crown on a posterior tooth. Each subject will use each of the study dentrifices over 3 months according to a randomization scheme. Subjects will brush daily with the assigned dentrifice unsupervised. Subjects will each have two provisonal crowns for use during the study. These crowns will contain three hard tooth tissue sections located at interproximal sites. The three tooth tissue slabs will consist of an artificial enamel caries lesion, an artificial root caries lesion, and a sound root. After removal, the tooth slabs will be evaluated using polarized light and photomicrographs for changes in area and depth of lesions.

ELIGIBILITY:
Inclusion Criteria:

* generally good physical health
* at least 18 years old
* needs a full crown on a mandibular first or second molar tooth
* tooth brushing frequency of twice daily or more
* agrees not to participate in other clinical study for duration of this study
* agrees to delay any elective dentistry, including dental prophylaxis, until study complete

Exclusion Criteria:

* any condition requiring antibiotic premedication before a dental procedure
* active treatment for cancer or seizure disorder
* diseases or conditions that could interfere with subject safely completing the study
* currently taking antibiotics or anti-cholinergic medications
* currently using extensive daily fluoride therapy
* gross, visible caries
* chronic use of chlorhexidine within 3 months of baseline
* use of systemic antibiotics within 7 days of baseline
* severe periodontal disease
* use of any fluoride rinses or gels one month prior to study initiation
* pregnancy, the intention to become pregnant
* presence of orthodontic bands or removable retainers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Generally healthy subjects in need of a full-coverage crown on a mandibular first or second molar
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in depth of artificial lesion over 3 months | 3 months
  Comparison of two 950 ppm fluoride containing dentrifices, Clinpro Toothcreme and MI Paste Plus, with fluoride-free dentrifice (Toms of Maine)for any change in artificial lesion depth due to demineralization or remineralization over the time period of the study
Change in area of artificial lesion over 3 months | 3 months
  Comparison of two 950 ppm fluoride containing dentrifices, Clinpro 5000 and MI Paste Plus, with fluoride-free dentrifice (Toms of Maine) for any change in artificial lesion area due to demineralization or remineralization over time period of study

CONTACTS AND LOCATIONS:
Overall Officials: Clark Stanford, PhD, Principal Investigator — Dows Institute for Dental Research
Locations (1):
- Dows Institute for Dental Research, Iowa City, Iowa, United States